CLINICAL TRIAL: NCT04064307
Title: Myotubular and Centronuclear Myopathy Patient Registry
Status: Recruiting | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: Myotubular Trust (Unknown); Muscular Dystrophy UK (Unknown); Astellas Gene Therapies (Industry); Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Chiara Marini Bettolo, Professor Neurologist and Clinical Lead, John Walton Muscular Dystrophy Research Centre. Clinical Lead of the Highly Specialised Service for Rare Neuromuscular Diseases, and Honorary Clinical Research Associate at Newcastle University, Newcastle-upon-Tyne Hospitals NHS Trust
Other Study IDs: NUTH 7729
Record Dates: First submitted 2018-03-06; First posted 2019-08-21 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Myotubular Myopathy; Myotubular Myopathy 1; Myotubular (Centronuclear) Myopathy; Centronuclear Myopathy; Centronuclear Myopathy, X-Linked; X-linked Myotubular Myopathy
Keywords: Registry; Patient Registry; Myotubular; Centronuclear; Myopathy
MeSH Terms: conditions — Myopathies, Structural, Congenital; Muscular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Myotubular and Centronuclear Myopathy Patient Registry (also referred to as the 'MTM and CNM Registry') is an international, patient-reported database specific to these conditions.

More details and online registration are available at www.mtmcnmregistry.org.

DETAILED DESCRIPTION:
The Myotubular and Centronuclear Myopathy (MTM & CNM) Patient Registry is managed and operated by the John Walton Muscular Dystrophy Research Centre at Newcastle University, in partnership with the Myotubular Trust, and is part of the TREAT-NMD Neuromuscular Network. The registry has been developed in partnership with a number of leading neuromuscular researchers, and is jointly funded by the Myotubular Trust, Muscular Dystrophy UK and Astellas Gene Therapies.

Participants register online and must provide consent before accessing the registry questionnaire. The clinical data and genetic or biopsy reports are provided by the participants and their doctors.

The MTM & CNM Registry aims to:

* Help identify patients for relevant clinical trials as they become available.
* Encourage further research into myotubular and centronuclear myopathy.
* Provide researchers with specific patient information to support their research.
* Assist doctors and other health professionals by providing them with up-to-date information on managing myotubular and centronuclear myopathy, to help them deliver better standards of care for their patients.

The investigators welcome the registration of:

* All patients with a myotubular myopathy or centronuclear myopathy diagnosis, which has been confirmed via genetic testing or muscle biopsy.
* Any carrier females of x-linked myotubular myopathy, especially if they have manifested myotubular myopathy type symptoms.
* Any patient who is deceased, but who had a confirmed diagnosis.

This is an online registry and is hosted on the RDRF (Rare Disease Registry Framework) by Murdoch University.

More details and online registration are available at www.mtmcnmregistry.org.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a myotubular myopathy or centronuclear myopathy diagnosis, which has been confirmed via genetic testing or muscle biopsy.
* Any carrier females of x-linked myotubular myopathy, especially if they have manifested myotubular myopathy type symptoms.
* Any patient who is deceased, but who had a confirmed diagnosis.

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible participants from any country. Registration is voluntary, and initiated by participants.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-03-26 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Patient questionnaire | 12 months
  Patient reported clinical diagnosis, genetic mutation, motor function, wheelchair use, respiratory function, ventilation type, chest infection, feeding and heart function, neuromuscular examinations, scoliosis surgery, family history and other registries joined. No scales are collected. Patient genetic report and muscle biopsy report are also uploaded to the registry if available, with details of clinician and where the tests were conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Marini Bettolo, Principal Investigator — Newcastle-upon-Tyne Hospitals NHS Trust
Locations (1):
- Newcastle University, Newcastle upon Tyne, Tyne and Wear, United Kingdom